CLINICAL TRIAL: NCT06298487
Title: Evaluation of the Multidimensional Impact of Therapeutic Education Workshops for COPD Patients, Cared for by the Maison de Prévention de la Santé et d'Accompagnement Thérapeutique, in the North-West Val d'Oise Area
Brief Title: Evaluation of the Impact of Therapeutic Education Workshops for COPD Patients in the North-West Val d'Oise Area
Acronym: MPSAT-ETP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There is no longer any point in continuing the research, as the objectives and evaluation criteria defined in the protocol are now being evaluated in everyday practice.
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHRD 1023
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-08

CONDITIONS: COPD
Keywords: COPD; Patient Therapeutic Education (PTE); House of Prevention-Health and Therapeutic Support (MPSAT); City-hospital
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTE group (Other): Group composed of patients who have already taken part in at least 3 Patient Therapeutic Education (PTE) workshops at the Maison de Prévention de la Santé et d'Accompagnement Therapeutique (MPSAT)
  Interventions: Other: Patient questionnaires
- Control group (Other): Group made up of patients on the waiting list for Patient Therapeutic Education (PTE) workshops at the Maison de Prévention de la Santé et d'Accompagnement Thérapeutique (MPSAT)
  Interventions: Other: Patient questionnaires

INTERVENTIONS:
Other: Patient questionnaires — Patients questionnaires, on paper or online (Microsoft Form) and data collection on patients medical file

SUMMARY:
The aim of this study is to assess the impact of the Patient Therapeutic Education (PTE) workshops offered by the Maison de Prévention de la Santé et d'Accompagnement Thérapeutique (MPSAT) on the follow-up and feelings of the COPD patients who take part. These workshops are organised outside the hospital environment and supervised by hospital and town professionals in the NOVO zone.

DETAILED DESCRIPTION:
In France, the ageing of the population (around 20% of the population is aged 65 or over), coupled with medical advances, lifestyle changes and environmental problems, is leading to an increase in chronic diseases, which are responsible for the majority of deaths.

Chronic obstructive pulmonary disease (COPD) is one of the most widespread chronic diseases in France. The departments most affected by COPD in terms of prevalence and (underestimated) mortality are the most vulnerable: Seine-et-Marne (77), Val-d'Oise (95) and Seine-Saint-Denis (93).

In the field of nursing, patient therapeutic education workshops (PTE) are an approach that aims to improve patients' health and well-being by actively involving them in managing their own health. The Maison de Prévention de la Santé et d'Accompagnement Thérapeutique (MPSAT), an innovative structure, seeks to promote this new approach by improving the management and care of COPD patients. In this context of changes in the management of the care pathway for chronic patients, one of the essential actions is therefore to actively involve the patient in the follow-up and to provide them with the means to understand their pathology: the main focus of this work will be on this crucial stage which is Patient Therapeutic Education (PTE). However, in 80% of cases, PTE programmes are developed almost exclusively in public hospitals. The PTE workshops run by the MPSAT, which take place outside the hospital, are fully justified here. The MPSAT, that will be at the heart of this research project, aims to promote this new approach by improving the management and care pathway for COPD patients.

The aim of this study is to answer the following question : in the context of developments in the management of patients suffering from chronic diseases in France, and in particular COPD, what is the impact of the MPSAT's therapeutic education workshops, organised outside the hospital environment and supervised by professionals from both the hospital and urban environments of the NOVO territory, on the COPD patients who take part in them?

ELIGIBILITY:
Inclusion Criteria :

* Patient aged 18 or over
* Patient living in the NOVO hospital area and the border towns of Yvelines, Oise and Eure
* Patient with a diagnosis of COPD confirmed by EFR, whatever the stage

For PTE group :

- Patient who has already attended at least 3 PTE workshops offered by MPSAT

For Control group :

- Patient on waiting list for PTE workshops offered by MPSAT

Exclusion Criteria :

* Patient refusing to take part in study
* Patient under legal protection
* Patient with cognitive disorders, unstable clinical conditions, language barriers or other conditions that prevent them from understanding the study and answering the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the overall impact of the PTE workshops offered by the MPSAT on patients' knowledge, skills, attitudes and behaviours with regard to COPD management and care | At the end of the study, an average of 6 month
  The overall impact of the PTE workshops will be assessed using the overall score of the HEIQ (Health Education Impact Questionnaire) validated in French It will be compared between patients in the PTE group (who attended at least 3 PTE workshops) and those in the control group (who did not attend any PTE workshops) For each item, the patient ticks the answer that best correspond to him or her : Strongly disagree, Disagree, Agree or Strongly agree

SECONDARY OUTCOMES:
Measure of the impact of PTE workshops on quality of life (comparison of PTE group versus Control group) | At the end of the study, an average of 6 month
  Patients' quality of life will be assessed using the validated short health-related quality of life questionnaire for routine practice in COPD patients (VQ11) and will be compared between both groups For each item, the patient ticks the answer that best correspond to him or her : Not at all, Somewhat, Moderately, Very much or Extremely
Comparison of anxiety/depression levels in patients in the PTE group versus Control group | At the end of the study, an average of 6 month
  Patients' anxiety and depression levels will be assessed using the validated Hospital Anxiety and Depression (HAD) questionnaire and will be compared between both groups For each item, the patient ticks the answer that best correspond to him or her with score between 0 and 3 (0 is the worst score and 3 the best score)
Comparison of levels of motivation towards physical activity during free time in the PTE group versus Control group | At the end of the study, an average of 6 month
  Motivation for physical activity during free time will be assessed using the short version of the questionnaire Behavioural Regulation in Exercise Questionnaire (BREQ-2) and will be compared between both groups the patient ticks the answer that best correspond to him or her :not at all true, moderately true or completely true
Comparison of the number of hospital admissions for COPD exacerbations in patients in the PTE group versus Control group | At the end of the study, an average of 6 month
  The number of hospitalisations of patients of PTE and Control groups will be obtained by examining their medical records and using the questionnaire on patient characteristics, which will provide information on any hospitalisations outside the NOVO hospital One of the questions in the questionnaire on patient characteristics concerns the number of hospitalisations, the year, the duration in days and the place of hospitalisation. For each item, the patient the patient can reply in free text
Comparison of the perception/feelings of patients in the PTE group versus Control group, concerning PTE workshops organised in a city/hospital setting | At the end of the study, an average of 6 month
  The workshops are offered close to home and run by two types of professional, one from the town and one from the hospital, with the possibility of integrating a new healthcare professional such as an advanced practice nurse The perception/feelings of patients in the PTE group versus Control group, regarding these workshops, will be evaluated using a questionnaire on patient follow-up and satisfaction For each question, the patient ticks the answer or answers that best correspond to him or her

CONTACTS AND LOCATIONS:
Overall Officials: Dr Bruno PHILIPPE, Principal Investigator — Hôpital NOVO
Locations (1):
- Pneumology, respiratory rehabilitation and follow-up and rehabilitation care department - Hôpital NOVO, Pontoise, France

REFERENCES:
- [Background] Adeloye D, Song P, Zhu Y, Campbell H, Sheikh A, Rudan I; NIHR RESPIRE Global Respiratory Health Unit. Global, regional, and national prevalence of, and risk factors for, chronic obstructive pulmonary disease (COPD) in 2019: a systematic review and modelling analysis. Lancet Respir Med. 2022 May;10(5):447-458. doi: 10.1016/S2213-2600(21)00511-7. Epub 2022 Mar 10. PMID 35279265
- [Background] Fuhrman C, Delmas MC; pour le groupe epidemiologie et recherche clinique de la SPLF. [Epidemiology of chronic obstructive pulmonary disease in France]. Rev Mal Respir. 2010 Feb;27(2):160-8. doi: 10.1016/j.rmr.2009.08.003. Epub 2010 Jan 19. French. PMID 20206064
- [Background] Brinchault G, Diot P, Dixmier A, Goupil F, Guillais P, Gut-Gobert C, Leroyer C, Marchand-Adam S, Meurice JC, Morel H, Person C, Cavailles A. [Comorbidities of COPD]. Rev Pneumol Clin. 2015 Dec;71(6):342-9. doi: 10.1016/j.pneumo.2015.09.009. Epub 2015 Nov 14. French. PMID 26585876
- [Background] Roche N, Zureik M, Soussan D, Neukirch F, Perrotin D; Urgence BPCO (COPD Emergency) Scientific Committee. Predictors of outcomes in COPD exacerbation cases presenting to the emergency department. Eur Respir J. 2008 Oct;32(4):953-61. doi: 10.1183/09031936.00129507. Epub 2008 May 28. PMID 18508819
- [Background] Bourbeau J, Julien M, Maltais F, Rouleau M, Beaupre A, Begin R, Renzi P, Nault D, Borycki E, Schwartzman K, Singh R, Collet JP; Chronic Obstructive Pulmonary Disease axis of the Respiratory Network Fonds de la Recherche en Sante du Quebec. Reduction of hospital utilization in patients with chronic obstructive pulmonary disease: a disease-specific self-management intervention. Arch Intern Med. 2003 Mar 10;163(5):585-91. doi: 10.1001/archinte.163.5.585. PMID 12622605
- [Background] Peytremann-Bridevaux I, Staeger P, Bridevaux PO, Ghali WA, Burnand B. Effectiveness of chronic obstructive pulmonary disease-management programs: systematic review and meta-analysis. Am J Med. 2008 May;121(5):433-443.e4. doi: 10.1016/j.amjmed.2008.02.009. PMID 18456040
- [Background] Bischoff EW, Hamd DH, Sedeno M, Benedetti A, Schermer TR, Bernard S, Maltais F, Bourbeau J. Effects of written action plan adherence on COPD exacerbation recovery. Thorax. 2011 Jan;66(1):26-31. doi: 10.1136/thx.2009.127621. Epub 2010 Oct 30. PMID 21037270
- [Background] Belanger A, Hudon C, Fortin M, Amirall J, Bouhali T, Chouinard MC. Validation of a French-language version of the health education impact Questionnaire (heiQ) among chronic disease patients seen in primary care: a cross-sectional study. Health Qual Life Outcomes. 2015 May 24;13:64. doi: 10.1186/s12955-015-0254-0. PMID 26306793